CLINICAL TRIAL: NCT05393661
Title: Implementation of Focused Intensive Repeated Stepping Training (FIRST) During Inpatient Rehabilitation Poststroke - A Quality Improvement Project
Brief Title: Focused Intensive Repeated Stepping During Inpatient Rehabilitation Poststroke - A Quality Improvement Project
Acronym: FIRST-IN
Status: Recruiting | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: ACL Administration for Community Living (Unknown); Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, George Hornby, Professor of Physical Medicine and Rehab, Indiana University
Other Study IDs: 1608161738
Record Dates: First submitted 2022-05-16; First posted 2022-05-26 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Stroke, Acute; Gait, Hemiplegic
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing inpatient rehabilitation poststroke: Inpatient rehabilitation poststroke
  Interventions: Other: inpatient physical therapy poststroke

INTERVENTIONS:
Other: inpatient physical therapy poststroke — routine care

SUMMARY:
The purpose of this quality improvement project was first to monitor usual physical therapy care (types & cardiovascular intensity of interventions and amount of stepping practice provided) and outcomes. Following which educational training and support was provided to treating physical therapists to encourage implementation of evidence-based practices. Specifically, therapists were encouraged to prioritize the practice of walking, particularly at higher cardiovascular intensities during scheduled therapy sessions. Fidelity metrics in the form of chart audits and pedometer-based step counts were utilized to determine compliance with the evidence-based intervention and ultimately investigated for potential effects on patient outcome measures.

DETAILED DESCRIPTION:
Converging data over the past 20 years suggest that the provision of large amounts of walking practice can improve walking function for individuals poststroke with greater improvements observed when the walking training is performed at moderate to high aerobic intensities. Despite this, current physical therapy practice during inpatient rehabilitation suggests limited walking practice is provided and low cardiovascular intensities achieved.

The purpose of this current quality improvement project is to evaluate the feasibility of implementing Focused, Intensive, Repeated Stepping Training (FIRST) during routine inpatient physical therapy and potential effects on patient outcome measures.

Prior to the usual care phase of the project, the outcome measures team worked to standardize routine collection of specific outcome measures (10 meter walk test, 6 minute walk test, Berg Balance Scale) at regular intervals (admission, weekly, discharge) in addition to 3rd party payer mandated measures (e.g., Functional Independence Measure; FIM). After which, existing physical therapy practice and outcomes will be monitored for a period of approximately 9-12 months. After which, educational training will be provided to physical therapists associated with the management of these patients as well as ongoing support (e.g., didactic, psychomotor, technical) and audit/feedback (e.g., chart audits, step count feedback) with fidelity metrics monitored from chart audits (walking practiced, walking prioritized, cardiovascular intensity documented, target intensity achieved) and pedometer step counts.

Potential changes in locomotor (e.g., 10 meter walk test, 6 minute walk test), non-locomotor outcomes (Berg Balance Scale, FIM-bed to chair transfers, FIM - toilet transfers), and incidence of adverse events will be evaluated if fidelity metrics indicate meaningful changes in clinical practice patterns. It is currently unknown what values of the fidelity metrics indicate successful implementation of the FIRST intervention, what knowledge translation strategies may be most effective to yield changes in therapists practice patterns, or the duration of time necessary to sufficiently achieve these changes in practice.

ELIGIBILITY:
Inclusion Criteria:

* < 2 months poststroke

Exclusion Criteria:

* restrictions in lower extremity weightbearing (e.g., amputation or lower limb fracture)
* unable to ambulate > 50 m prior to their most recent stroke
* discharged to home from inpatient rehabilitation after < 1 week

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals admitted to the Rehabilitation Hospital of Indiana for acute inpatient rehabilitation poststroke
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in 10 meter walk test | Time from admission & discharge inpatient rehabilitation or approximately 20 days
  Differences in time for individual to ambulate 10 meters (with middle 6 meters timed) with directions "walk at your usual, comfortable pace" from admission and discharge from inpatient rehabilitation
Change in 6 minute walk test | Time from admission & discharge inpatient rehabilitation or approximately 20 days
  Differences in distance able to be ambulated during a 6 minute period with directions "cover as much ground as possible" from admission and discharge from inpatient rehabilitation
Change in 6 minute walk test level of assistance | Time from admission & discharge inpatient rehabilitation or approximately 20 days
  Differences in amount of physical assistance provided by physical therapist during 6 minute walk test

SECONDARY OUTCOMES:
Change in Berg Balance Scale | Time from admission & discharge inpatient rehabilitation or approximately 20 days
  Differences in performance on a 14 item static balance assessment
Change in Functional Independence Measure - bed to chair transfer subscore | Time from admission & discharge inpatient rehabilitation or approximately 20 days
  Differences in performance during task assessed using an ordinal score (0-7) for amount of physical assistance necessary to complete functional task
Change in Functional Independence Measure - toilet transfer subscore | Time from admission & discharge inpatient rehabilitation or approximately 20 days
  Differences in performance during task assessed using an ordinal score (0-7) for amount of physical assistance necessary to complete functional task
Change in Functional Independence Measure - locomotion | Time from admission & discharge inpatient rehabilitation or approximately 20 days
  Differences in performance during task assessed using an ordinal score (0-7) for amount of physical assistance necessary and distance covered during level overground ambulation
Change in Functional Independence Measure - stairs | Time from admission & discharge inpatient rehabilitation or approximately 20 days
  Differences in performance during task assessed using an ordinal score (0-7) for amount of physical assistance necessary and number of stairs able to be negotiated

OTHER OUTCOMES:
Incidence of significant adverse events | Throughout time from admission & discharge inpatient rehabilitation or approximately 20 days
  Includes death, new cerebrovascular events, or rehospitalization
Incidence of falls without injuries | Throughout time from admission & discharge inpatient rehabilitation or approximately 20 days
  Medical documentation indicating a fall without an associated significant adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Hornby, Principal Investigator — Indiana University
Locations (1):
- Rehabilitation Hospital of Indiana, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data available upon reasonable request
Time Frame: after completion of study for 3 years